CLINICAL TRIAL: NCT04101097
Title: Training and Validation of Models Based on Patient-related or Procedure-related Factors to Predict Inadequate Bowel Preparation in Patients Undergoing Colonoscopy
Brief Title: Training and Validation of Models of Factors to Predict Inadequate Bowel Preparation Colonoscopy
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other); Xiamen Humanity Hospital (Other); Huaihe Hospital of Henan University (Other); Shaanxi Second People's Hospital (Unknown)
Responsible Party: Principal Investigator, Yanglin Pan, Associate Professor, Air Force Military Medical University, China
Other Study IDs: KY20190903-3
Record Dates: First submitted 2019-09-21; First posted 2019-09-24 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Colonoscopy; Bowel Preparation; Predictive Model
Keywords: factors;bowel preparation;colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training group: All patients received oral and written instructions on the appointment day. All patients were instructed to have low-residue food for lunch and dinner on the day before colonoscopy. Patients were instructed to begin drinking the first 1.5L-2L PEG at 7:00-9:00 PM on the day before colonoscopy. On the day of the procedure, they took another 1.5L-2L 4-6 hours before colonoscopy. Patients were encouraged more to drink more clear liquids after purgatives for adequate hydration.
- validation group: All patients received oral and written instructions on the appointment day. All patients were instructed to have low-residue food for lunch and dinner on the day before colonoscopy. Patients were instructed to begin drinking the first 1.5L-2L PEG at 7:00-9:00 PM on the day before colonoscopy. On the day of the procedure, they took another 1.5L-2L 4-6 hours before colonoscopy. Patients were encouraged more to drink more clear liquids after purgatives for adequate hydration.

INTERVENTIONS:
Other:

SUMMARY:
The rate of adequate bowel preparation is one of important quality indicators of colonoscopy. Inadeqaute bowel preparation negatively affects the outcomes of colonoscopy. If patients with inadequate bowel preparation were identified before the procedure, enhanced strategy could be offerred to achieve better bowel cleasing. Currently, there were three predicting models of inadequate bowel preparation eatablished based on patient-related factors. It remains unclear which model perfroms better in predicting bowel preparation quality. Futhermore, althought those predicting models only composing of patients-related factors are useful for identifing high-risk patients, the preparation-related factors may also be valuable for prediciting inadeqaute bowel preparation before the procedure of colonoscopy.

This study aimed: 1) to compare the values of three availlable models (based on patient-related factors) in predicting inadeqaute bowel preparation in a prospective, multicentered cohort of patients undergoing colonoscopy; 2) to investigate whether a new model based on preparation-related or a combined model based on patient-related and preparation-related factors is comparable to previous models based on patient-related factors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80
* Using PEG for bowel preparation before colonoscopy

Exclusion Criteria:

* Not undergoing standard bowel preparation due to emergency, bleeding or unsuitable for preparation
* Colon resection
* Suspected bowel obstruction
* Hemodynamically unstable
* Lactating or pregnant women
* Unwilling to provided informed content

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using PEG for bowel preparation before colonoscopy
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Inadequate bowel preparation | 1 hour
  Inadequate bowel preparation was defined by the Boston Bowel Preparation Scale of any segmental<2.

SECONDARY OUTCOMES:
Adequacy of proximal bowel preparation | 1 hour
  Adequate bowel preparation is defined by the Boston Bowel Preparation Scale of right-colon<2 or middle colon<2
Adequacy of distal bowel preparation | 1 hour
  Adequate bowel preparation is defined by the Boston Bowel Preparation Scale of left-colon<2 or middle colon<2

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Department of Gastroenterology, Hongai Hospital, Xiamen, Fujian
  - Department of Holistic Integrative Medicine, Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Department of Gastroenterology, Huaihe Hospital of Henan University, Kaifeng, Henan
  - Department of Gastroenterology, Shaanxi Second People's Hospital, Xi'an, Shaanxi
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi

REFERENCES:
- [Result] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Result] Dik VK, Moons LM, Huyuk M, van der Schaar P, de Vos Tot Nederveen Cappel WH, Ter Borg PC, Meijssen MA, Ouwendijk RJ, Le Fevre DM, Stouten M, van der Galien O, Hiemstra TJ, Monkelbaan JF, van Oijen MG, Siersema PD; Colonoscopy Quality Initiative. Predicting inadequate bowel preparation for colonoscopy in participants receiving split-dose bowel preparation: development and validation of a prediction score. Gastrointest Endosc. 2015 Mar;81(3):665-72. doi: 10.1016/j.gie.2014.09.066. Epub 2015 Jan 17. PMID 25600879
- [Result] Gimeno-Garcia AZ, Baute JL, Hernandez G, Morales D, Gonzalez-Perez CD, Nicolas-Perez D, Alarcon-Fernandez O, Jimenez A, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Carrillo M, Ramos L, Quintero E. Risk factors for inadequate bowel preparation: a validated predictive score. Endoscopy. 2017 Jun;49(6):536-543. doi: 10.1055/s-0043-101683. Epub 2017 Mar 10. PMID 28282690